CLINICAL TRIAL: NCT03819361
Title: Effect of Longitudinal Sleep Monitoring on Diagnosis and Treatment Decision in Patients with Suspected Obstructive Sleep Apnea (ELSA)
Brief Title: Effect of Longitudinal Sleep Monitoring on Diagnosis and Treatment Decision in Patients with Suspected Obstructive Sleep Apnea
Acronym: ELSA
Status: Active, not recruiting | Type: Observational
Sponsor: Malcolm Kohler (Other)
Responsible Party: Sponsor-Investigator, Malcolm Kohler, Head of the department of pulmonology, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2018-02305
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Night-to-night variability; Apnoea-Hypopnoea Index; Oxygen Desaturation Index; Pulse-oximetry
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Suspected OSA
  Interventions: Diagnostic Test: pulse-oximetry

INTERVENTIONS:
Diagnostic Test: pulse-oximetry — Patients with suspected OSA will be monitored with 14 nights of pulse-oximetry prior to the already planned in-hospital single-night sleep study at the University Hospital Zurich

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent sleep-disordered breathing disease, caused by recurrent episodes of partial or complete collapse of the upper airway during sleep, resulting in intermittent hypoxia, fragmented sleep, fluctuations in blood pressure, and increased sympathetic nervous system activity. A single-night sleep study (i.e. respiratory polygraphy or polysomnography) is currently considered to be the gold standard for diagnosing OSA. However, recent studies suggest a significant intra-individual night-to-night variability of respiratory events, leading to the hypothesis that one single-night study might not reflect an accurate picture of the disease.

Part A: Patients with suspected obstructive sleep apnea, referred to our clinic, undergo the regular diagnostic procedure recommended by the current guidelines. In addition to the in-hospital single-night sleep study, these patients will perform 14 nights of pulse-oximetry at home. By computing and analysing sensitivity and specificity of every additional night, the investigator will answer the questions how many nights of sleep monitoring by home oximetry are necessary to diagnose OSA reliably, and how longitudinal sleep monitoring could reduce the number of false-negative and false- positive results compared to the in-hospital single-night study.

Part B: Based on the patients' data of part A, the investigator will develop a questionnaire and present anonymized cases to experts in the field of sleep medicine. Thereby, the investigator will evaluate if the additional information of repeated nocturnal pulse-oximetries changes the experts' decision making regarding diagnosis and treatment of OSA.

In a second step, the investigator will perform a classical Delphi study with a panel of experts in sleep medicine to establish consensus on repeated sleep studies and how they should be used for diagnosis and treatment in patients with suspected OSA.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Suspected obstructive sleep apnea
* ≥18 years old

Exclusion Criteria:

* Suspected or diagnosed sleeping-disordered breathing other than OSA
* Moribund or severe disease prohibiting protocol adherence especially COPD GOLD III-IV and heart failure NYHA III-IV
* Patients receiving oxygen therapy or home ventilation
* Continuous positive airway pressure treatment for OSA at baseline
* Physical or intellectual impairment precluding informed consent or protocol adherence
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with suspected obstructive sleep apnea
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of 1-13 nights of pulse-oximetry compared to the mean ODI of 14 consecutive nights | 14 nights of pulse-oximetry
  "Sensitivity" and "specificity" for every additional night will be assessed
Decision making of a panel of experts in the field of sleep medicine regarding diagnosis and severity of OSA (no OSA, mild, moderate, severe) with/without the additional information of longitudinal sleep monitoring | 14 nights of pulse-oximetry

SECONDARY OUTCOMES:
ODI variability measured in 14 consecutive nights of pulse-oximetry | 14 nights of pulse-oximetry
Change of OSA severity class (no OSA, mild, moderate, severe OSA) during 14 nights of pulse-oximetry due to ODI variability | 14 nights of pulse-oximetry
Change of OSA severity class (no OSA, mild, moderate, severe OSA) diagnosed by in-hospital single-night sleep study vs repeated measurements by pulse-oximetry | 14 nights of pulse-oximetry
Decision making of a panel of experts in field of sleep medicine regarding treatment decisions (CPAP yes/no) with/without the additional information of longitudinal sleep monitoring | 14 nights of pulse-oximetry
Establish consensus on repeated sleep studies and their use in diagnosis and treatment in patients with suspected OSA | 14 nights of pulse-oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, Prof. Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roeder M, Sievi NA, Bradicich M, Grewe FA, Siegfried S, Gaisl T, Kohler M. The Accuracy of Repeated Sleep Studies in OSA: A Longitudinal Observational Study With 14 Nights of Oxygen Saturation Monitoring. Chest. 2021 Mar;159(3):1222-1231. doi: 10.1016/j.chest.2020.09.098. Epub 2020 Sep 25. PMID 32980370